CLINICAL TRIAL: NCT04115592
Title: The Effect of Different States of Lipid in Food on Glycaemia, Lipaemia and Insulinaemia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2018/01193
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Risk Factor
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — cocoa butter

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Liquid oil type 1 (Experimental): Cocoa butter (CB)
  Interventions: Other: Cocoa butter
- Solid oil type 1 (Experimental): Cocoa butter oleogel (CBOG)
  Interventions: Other: Cocoa butter oleogel
- Liquid oil type 2 (Experimental): Sal seed oil (SL)
  Interventions: Other: Sal seed oil
- Solid oil type 2 (Experimental): Sal seed oleogel (SLOG)
  Interventions: Other: Sal seed oleogel

INTERVENTIONS:
Other: Cocoa butter — Consumption of cocoa butter made with chocolate confectionery
  Arms: Liquid oil type 1
Other: Cocoa butter oleogel — Consumption of cocoa butter oleogel made with chocolate confectionery
  Arms: Solid oil type 1
Other: Sal seed oil — Consumption of sal seed oil made with chocolate confectionery
  Arms: Liquid oil type 2
Other: Sal seed oleogel — Consumption of sal seed oleogel made with chocolate confectionery
  Arms: Solid oil type 2

SUMMARY:
The aim of this study is to investigate if the application of lipid in various form (i.e. liquid and solid) affects glycaemia, lipaemia and insulinaemia. In addition, this study aims to test the lipidemic effects of the use of vegetable oil as a substitute in the application for making chocolate confectionery.

DETAILED DESCRIPTION:
The study will have a randomized, non-blinded, crossover design. This study will explicitly compare the effects of different forms of fat (liquid and solid) on glucose, insulin and lipid response on 20 healthy male participants between the age of 21-40 years. In addition, this study aims to test the lipidemic effects of the use of vegetable oil as a substitute in the application for making chocolate confectionery.

All potential participants will be asked to attend four testing sessions and a screening session in total. During the first screening session, participants will receive an informed consent form and given ample time to go through it and rectify any queries they have. If they decide to take part in the study, they will be asked to sign the informed consent form. They will then be asked to complete a screening questionnaire, baseline measurements including anthropometric measurements, blood pressure, and fasting blood glucose will be collected from each participant in order to determine their eligibility. During the test sessions, participants' glycaemic, insulinaemic and lipaemic responses to the test meals will be measured. The test duration for each session will be 6.5 hours. Participants will be instructed to avoid strenuous physical activity for at least 3 days and avoid caffeine and alcohol consumption for at least 1 day prior to visiting the CNRC for their study trials. Participants will be provided with a standardized dinner meal (consisting of rice/noodles, vegetables, meat, drink/pudding) and to refrain from alcohol and exercise the day before their testing sessions.

Screening questionnaire: The screening questionnaire will include contact information, demographic and general health details. This information will be used to determine whether the participant is eligible for the study, as well as to check for any possible confounders that may influence the study outcomes.

Anthropometric measurements: Body weight and body composition will be measured using bioelectrical impedance analysis. Height will be measured using a stadiometer in order to calculate participants' BMI. Blood pressure will also be measured. All measurements will be taken in duplicate during the screening session. Waist circumference will be measured at the minimum circumference between the iliac crest and the rib cage. Hip circumference will be measured at the maximum protuberance of the buttocks. Biceps and triceps skinfold measurements will also be taken. Blood pressure will be measured using an Omron blood pressure monitor (Model HEM-907) at baseline. Participants will be seated for five minutes before blood pressure is measured. Measurements will be taken in duplicate and the averaged results will be recorded.

Blood collection: Participants will be asked to attend the testing sessions after an overnight fast of ten hours. At the beginning of the testing session, a cannula will be inserted into participants' arms. One fasting blood sample will be collected by venous cannulation. 3 milliliters (ml) of venous blood will be collected into Vacutainers® (Belton Dickinson Diagnostics) containing disodium EDTA for the analyses of plasma triglyceride, glucose and insulin concentrations. Participants will then consume treatment meal within 15 minutes. Blood samples will be taken at baseline, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330 and 360 minutes. The amount of blood that will be collected at every time point will be approximately 3ml. A maximum of 15 blood samples will be collected by cannulation. A total of 180ml of blood will be taken for the study. Glycaemic, insulinaemic, and lipaemic responses will be determined using the method described by Wolever and Jenkins. The area under the curve will be determined as the area of those increments above baseline only.

Test session: Participants will be provided a standard dinner meal to be consumed at home at 7pm the night before the test session. Afterwhich, they will be asked to not eat and drink anything except water after 10:30 pm. They will also be instructed to arrive at the CNRC the following morning after an overnight fast of 10-12 hours. After 10 minutes upon arrival, an indwelling catheter will be inserted into a vein in your forearm and will be kept patent (free of clots) for the remainder of the test session. We will then take a blood sample from the cannula to measure baseline values. After obtaining the baseline blood samples, participants will be given the test meal to consume within 15 minutes. Following the test meal, we will take further blood samples (from the cannula) for the next 15, 30, 45, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 360 minutes. The cannula will be removed after the last time-point of blood sample collection (360 minutes) and they are free to leave CNRC. During the entire testing period the participants will be instructed to remain rested and in the laboratory. There will be no incidental findings as analysed samples are basic metabolites and therefore, reporting is not applicable.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Healthy Asian Chinese
* Aged between 21 - 40 years
* ≥45kg body weight
* Body mass index between 18.5 to 25.0 kg/m2
* Normal blood pressure ≤140/90 mmHg
* Fasting blood glucose <5.6 mmol/L

Exclusion Criteria:

* Smoking
* Allergic/intolerant to any of the test foods to be administered, or any of the following common food and ingredients: eggs, fish, milk, peanuts, and tree nuts, shellfish, soya, wheat, gluten, cereal, fruits, dairy products, meat, vegetable, sugar and sweetener, natural food colourings or flavourings, etc.
* Anyone with intentional food restrictions
* People with known glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Having metabolic or cardiovascular diseases (such as diabetes, hypertension, heart condition, etc.), Having any other diseases involving the small intestine or the colon (e.g., irritable bowel syndrome, inflammatory bowel disease, gastric reflux) or having any liver or kidney disorders or any family history of kidney stones
* Having medical conditions and/or taking medications known to affect glycaemia (glucocorticoids, thyroid hormones, thiazide diuretics)
* Taking any prescribed medication or dietary supplements which may interfere with the study measurements
* Individuals who have any major organ dysfunction (eg. cardiovascular, respiratory, hepatic, renal, gastrointestinal) that may influence taste, olfaction, appetite, digestion, metabolism, absorption or elimination of test foods, nutraceutical or drug
* Excessive alcohol consumption: consuming ≥ 6 alcoholic drinks per week
* Have known Chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Have active Tuberculosis (TB) or currently receiving treatment for TB
* Individuals who partake in sports at the competitive and/or endurance levels
* A team member of the study or is an immediate family member (Immediate family defined as a spouse, parent, child, or sibling, whether biological or legally adopted

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All healthy male volunteers
Enrollment: 19 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Postprandial triglycerides | From 0 to 360 minutes
  Venous blood plasma measured using the COBAS
Postprandial glucose | From 0 to 360 minutes
  Venous blood plasma measured using the COBAS

SECONDARY OUTCOMES:
Postprandial insulin | From 0 to 360 minutes
  Venous blood plasma measured using the COBAS

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore